CLINICAL TRIAL: NCT01159119
Title: Single Center Randomized Single Blind Crossover Group Active Control Study to Evaluate Safety and Efficacy of EUR-1066 a Pancreatic Enzyme Product in Patients With Chronic Pancreatitis Exocrine Pancratic Insufficiency,Chronic Abdominal Pain
Brief Title: A Study of EUR-1066 in Subjects With Chronic Pancreatitis, Exocrine Pancreatic Insufficiency and Chronic Abdominal Pain
Acronym: EUR-1066
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PR-012
Record Dates: First submitted 2010-07-05; First posted 2010-07-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic Abdominal Pain; Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- EUR-1066-A (Experimental): Treatment with Eur-1006-A.
  Interventions: Drug: EUR-1066-A
- EUR-1066-B (Experimental): Treatment with Eur-1066-B
  Interventions: Drug: EUR-1066-B
- Zenpep (Active Comparator): Control Group: Consist of treatment with Zenpep
  Interventions: Drug: Zenpep

INTERVENTIONS:
Drug: EUR-1066-A — Eur-1066 capsules taken daily for 28 days either during treatment period 1 or treatment period 3.
  Other Names: EUR-1066
  Arms: EUR-1066-A
Drug: Zenpep — Capsules taken for daily for 28 days during treatment period 2
  Arms: Zenpep
Drug: EUR-1066-B — Eur-1066 capsules taken daily for 28 days either during treatment period 1 or treatment period 3.
  Other Names: EUR-1066
  Arms: EUR-1066-B

SUMMARY:
The purpose of this study is to evaluate two different treatments in subjects with chronic pancreatitis, exocrine pancreatic insufficiency and chronic abdominal pain.

DETAILED DESCRIPTION:
To evaluate two different preparations of a pancreatic enzyme in subjects with chronic pancreatitis, exocrine pancreatic insufficiency, and chronic abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Pancreatitis
* Exocrine Pancreatic Insufficiency
* Chronic abdominal pain

Exclusion Criteria:

* Acute pancreatitis
* Active alcohol consumption
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-08-02 (Actual); Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
Comparing frequency and severity of pain | up to 84 days
  Patient diary

SECONDARY OUTCOMES:
Changes in fat malabsorption | up to 124 days
  Assess the coefficient of fat absorption

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Toskes, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States